CLINICAL TRIAL: NCT06244641
Title: Creation of a Visualization Tool With Integrated Clinical Data to Support Clinical Intervention and Empowerment of Inpatients in Psychiatry : Basis for the Development of a Predictive Model of Relapse
Brief Title: New Relapse Model in Psychiatry
Acronym: NRMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/09MAI/22
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
Keywords: clustering; relapse; feedback-measurment-system
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Evoked Potentials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Auto-questionnaires, hetero-questionnaires and Evoked-potentials

INTERVENTIONS:
Other: Auto-questionnaires, hetero-questionnaires and Evoked-potentials — Evaluations of risk factors of relapse by questionnaires, evaluation of evoked-potentials

SUMMARY:
The goal of this clinical trial is to learn about risk factors of relapse in patients with alcohol use disorder. The main questions it aims to answer are :

* Among patients with Alcohol Use Disorder, are there clusters of patients with the same characteristics and the same outcome ?
* Which are the risk factors of relapse that are the most predictive ? Do they vary according to cluster?
* Can a feedback-measurment-system (eg : a feedback of the tests' results) be usefull in a detoxification unit ?

Participants will :

* Complete auto-questionnaires
* Pass hetero-evaluations
* Undergo an electrophysiological battery

ELIGIBILITY:
Inclusion Criteria:

* To suffer from AUD
* To be hospitalized
* To speak French fluently
* To be able to give their consent (medically and legally).

Exclusion Criteria:

* To suffer from severe perceptive disabilities (auditory, visual)
* To suffer from severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Relapse or abstinence after detoxification | Throughout the entire study, approximately during 48 months
  number of alcohol units and time to relapse or abstinence after detoxification

SECONDARY OUTCOMES:
Satisfaction of the feedback-measurment-system for clinicians and patients | Throughout the entire study, approximately during 48 months
  Simple questions with Likert-scale to evaluate the feedback-measurment-system

CONTACTS AND LOCATIONS:
Overall Officials: Philippe de Timary, PhD, Principal Investigator — Université catholique de Louvain (Wallonia)
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided